CLINICAL TRIAL: NCT04707872
Title: Trifecta-Heart cfDNA-MMDX Study: Comparing the DD-cfDNA Test to MMDx Microarray Test and Central HLA Antibody Test
Brief Title: Trifecta-Heart cfDNA-MMDx Study
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Natera, Inc. (Industry); One Lambda (Unknown)
Responsible Party: Sponsor
Other Study IDs: ATAGC06
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplant Rejection
Keywords: Donor derived cfDNA; gene expression; heart transplant biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — RNA isolated from patient biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart transplant protocol and for cause biopsies: The study population includes patients with a functioning heart transplant undergoing a biopsy for clinical indications as standard of care, or protocol biopsies of heart in high-risk patients, or follow-up after treatment.
  Interventions: Diagnostic Test: MMDx diagnostic test; Diagnostic Test: Prospera; Diagnostic Test: HLA antibody

INTERVENTIONS:
Diagnostic Test: MMDx diagnostic test — Microarray test of gene expression in heart biopsies
Diagnostic Test: Prospera — Donor derived cell-free DNA in patient blood
Diagnostic Test: HLA antibody — Centralized measurement of HLA antibodies in patient blood

SUMMARY:
Demonstrate the relationship between DD-cfDNA levels and HLA antibodies in blood transplant recipient and the Molecular Microscope® (MMDx) Diagnostic System results in indication and protocol biopsies from heart transplants.

DETAILED DESCRIPTION:
The current standard for assessment of rejection in heart transplants is an endomyocardial biopsy (EMB) interpreted by histology according to ISHLT guidelines. This has considerable error rates, many due to the high disagreement among pathologists in assessing lesions and diagnoses. To address the unmet need for precision and accuracy, the Alberta Transplant Applied Genomics Centre (ATAGC, University of Alberta) has developed a new diagnostic system - the Molecular Microscope® Diagnostic System (MMDx), which uses microarrays to define the global gene expression features of rejection and injury. Now a new screening test is being introduced: the monitoring of donor-derived cell-free DNA (DD-cfDNA) released in the blood by the heart during rejection. The Natera Inc DD-cfDNA Prospera® test is based on the massively multiplex polymerase chain reaction that targets 13,392 single nucleotide polymorphisms and targeted sequences are quantified by Next Generation Sequencing. The Prospera® test has been done on kidney transplant recipients and detected "active rejection" and differentiated it from borderline rejection and no rejection. However, Prospera® test was not examined (the DD-cfDNA results) in heart transplant recipients. DD-cf-DNA test for heart transplants must now be calibrated against MMDx that is based on global gene expression, the new standard for biopsy interpretation. The present study will calibrate centrally measured (Natera Inc) DD-cfDNA levels obtained at the time of an indication or protocol biopsy against the MMDx measurements of T cell-mediated rejection (TCMR), antibody-mediated rejection (ABMR) and early and late tissue injury. The present study will compare DD-cfDNA and MMDx in 300 prospectively collected biopsies for clinical indications and protocol, and accompanying 600 blood samples, to calibrate the DD-cfDNA (Natera Inc.) levels against the MMDx biopsy diagnoses of TCMR, ABMR (and its stages), and acute (early) and chronic (late) injury, , as well as central assessment of HLA antibody (One Lambda) in 300 blood samples, interpreted centrally as donor specific antibody (DSA) based on the tissue typing results. Trifecta-Heart collected 658 biopsies, 609 cfDNA samples and 640 One Lambda samples so far. Due to a considerable interest from participation centers, this study aims to collect 300 more biopsies and corresponding blood samples. This study is an extension of the INTERHEART ClinicalTrials.gov Identifier: NCT02670408

ELIGIBILITY:
Inclusion Criteria:

* All heart transplant recipients undergoing a biopsy for clinical indications and protocol biopsies, as determined by their physician or surgeon, will be eligible to enroll in the study.
* Patients are enrolled based on standard of care biopsies, including surveillance biopsies in high-risk patients, with informed consent.

Exclusion Criteria:

* Patients will be excluded from the study if they decline participation
* Are unable to give informed consent.
* Recipients of multiple organs.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes patients with a functioning heart transplant undergoing a biopsy for clinical indications or surveillance (protocol) biopsy.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Calibration of Prospera test for T cell-mediated rejection | 18 months
  Set DD-cfDNA test cut-off values against the probability of T cell-mediated rejection in the biopsy as reported by MMDx. Calibration of DD-cfDNA test cut-off values against the probability of T cell-mediated rejection in the biopsy as reported by MMDx.
Calibration of Prospera test for antibody-mediated rejection | 18 months
  Set DD-cfDNA test cut-off values against the probability of antibody-mediated rejection in the biopsy as reported by MMDx.
Calibration of Prospera test for heart injury | 18 month
  Set DD-cfDNA test cut-off values against the probability of acute and chronic heart injury in the biopsy as reported by MMDx.
Report calibrated Prospera test results for rejection | 6 months
  Obtain clinicians feedback
Report calibrated Prospera test results for heart injury | 6 month
  Obtain clinicians feedback

SECONDARY OUTCOMES:
Determine if Prospera blood test can replace heart biopsy test | 6 month
  Obtain clinicians feedback
Determine if Prospera blood test can replace follow up heart biopsy | 6 month
  Determine whether resolution of DD-cfDNA after treatment can monitor response to therapy and avoid follow-up biopsies
Assessment of donor-specific antibody status | 6 months
  Report and compare the DSA status based on centralized and local HLA antibody measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Philip F Halloran, MD PhD, Principal Investigator — Alberta Transplant Applied Genomics Center, University of Alberta
Locations (12):
- United States (6):
  - Baptist Health Institute for Research and Innovation, Little Rock, Arkansas
  - Tampa General Hospital, 409 Bayshore Blvd., Tampa, Florida
  - Columbia University Medical Center, Columbia Interventional Cardiovascular Care, West New York, New Jersey
  - Montefiore Medical Center, 3319 Rochambeau Avenue, 2nd FL, The Bronx, New York
  - Annette C. and Harold C. Simmons Transplant Institute, BaylorScott&White Research Institute, Dallas, Texas
  - Cardiovascular Medicine, University of Utah Health, Salt Lake City, Utah
- Cardiac Transplantation Laboratory, The Victor Chang Cardiac Research Institute, Darlinghurst, Australia
- Division of Cardiology, University of Alberta, Edmonton, Alberta, Canada
- Institute for Clinical and Experimental Medicine - IKEM Videnska 1958/9, Prague, Czechia
- Heart Failure and Heart Transplant Unit, University of Bologna, Bologna, Italy
- Silesian Center for Heart Diseases (Ś!ąskie Centrum Chorób Serca w Zabrzu, Zabrze, Poland
- Advanced Heart Failure Transplant Unit, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No
Only IPD data will be shared within a participating center.

REFERENCES:
- [Background] Madill-Thomsen KS, Halloran PF. Precision diagnostics in transplanted organs using microarray-assessed gene expression: concepts and technical methods of the Molecular Microscope(R) Diagnostic System (MMDx). Clin Sci (Lond). 2024 Jun 5;138(11):663-685. doi: 10.1042/CS20220530. PMID 38819301
- [Background] Halloran PF, Madill-Thomsen KS. Donor-derived Cell-free DNA: A Step Forward in the Quest for Transplant Truth. Transplantation. 2025 Jun 1;109(6):910-914. doi: 10.1097/TP.0000000000005332. Epub 2025 Jan 28. No abstract available. PMID 39883025
- [Result] Halloran PF, Reeve J, Mackova M, Madill-Thomsen KS, Demko Z, Olymbios M, Campbell P, Melenovsky V, Gong T, Hall S, Stehlik J. Comparing Plasma Donor-derived Cell-free DNA to Gene Expression in Endomyocardial Biopsies in the Trifecta-Heart Study. Transplantation. 2024 Sep 1;108(9):1931-1942. doi: 10.1097/TP.0000000000004986. Epub 2024 Aug 20. PMID 38538559
- [Result] Madill-Thomsen KS, Hidalgo LG, Mackova M, Campbell P, Demko Z, Felius J, Gong T, Hall S, Kim DH, Kuczaj A, Lowe D, Maliakkal N, Melenovsky V, Olympios M, Patel S, Prewett A, Przybylowski P, Sayer G, Stehlik J, Tseliou E, Uriel N, Halloran PF. Defining the relationships among four tests for assessing antibody-mediated rejection in heart transplants in a prospective, observational study. J Heart Lung Transplant. 2025 Nov 13:S1053-2498(25)02363-0. doi: 10.1016/j.healun.2025.10.024. Online ahead of print. PMID 41241034
- [Derived] Halloran PF, Madill-Thomsen KS. The Molecular Microscope Diagnostic System: Assessment of Rejection and Injury in Heart Transplant Biopsies. Transplantation. 2023 Jan 1;107(1):27-44. doi: 10.1097/TP.0000000000004323. Epub 2022 Dec 8. PMID 36508644